CLINICAL TRIAL: NCT03716882
Title: Acoustic Structures Crying of Infants From 1 to 4 Months and Their Signification
Acronym: LongCRY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: ENES, CNRS 9197 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18CH085; 2018-A01399-46 (Other: ANSM)
Record Dates: First submitted 2018-10-22; First posted 2018-10-23 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Infants
Keywords: Infants; Principal Component 1 (PC1); Principal Component 2 (PC2); Song Meter 4; Acoustic structures crying; PRAAT software

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infant at the birth: Infant at the birth will be included. Their cries will be longitudinally registered using an automatic record device: Song Meter (SM)4 during 3 consecutive days and nights.
  At every cry, parent should answer the questionnaire of cry in infant.
  Interventions: Device: Song Meter (SM)4

INTERVENTIONS:
Device: Song Meter (SM)4 — Their cries will be longitudinally registered using an automatic record device: Song Meter (SM)4 during 3 consecutive days and nights. This record will take place at 15 days of life, 1 and half months, 2 and half months and 3 and half months.
  Other Names: automatic record device

SUMMARY:
Crying is a survival mechanism for babies and their almost exclusive means of expression until the age of 4 months. Babies 'cry is mostly related to pain, a feeling of hunger, discomfort or separation following the departure of a parent around. Crying is a complex but essential means of communication and information between a baby and his parents that raises the question of their meaning.

The cry phenomenon consists of complex acoustic signals produced by the vocal cords and filtered by the vocal tract. The vibrations frequency determines the fundamental frequency, itself responsible for the perception of the cry tone (pitch). The frequency spectrum of a cry is modified during the passage through the upper airways forming broad bands called "resonance frequency" or "formants".

From the specificity of a crying sequence, it is possible to extract dynamic information and relate it to the perception that the adult has of it. Thus dynamic crying is often perceived by the adult as an imminent need of the baby.

Some studies have shown that a child's crying may change according to his degree of discomfort, suggesting that crying was a "graduated signal" whose frequency and timbre could vary along a continuum. These changes would explain why adult listeners would be able to dissociate crying babies of different intensities.

Conversely, an inappropriate response to crying could gradually generate disorders of the relationship between the baby and the parent.

However, despite their potential neuro-ethological interest, knowledge of information transmitted by babies's cry remains superficial. This could be related to the relatively obsolete techniques of recording or due to the lack of objective physiological data on babies 'cry. Finally, the perception and reactions of adults when they hear crying babies are not fully understood.

DETAILED DESCRIPTION:
The objective of this study is to evaluate acoustic structures crying of infants from 1 to 4 months for to study individual acoustic signature.

ELIGIBILITY:
Inclusion Criteria:

* any safe term infants (> 37SA)
* eutrophic and in good health
* infants sleeping in bed with bars without baby nest
* form signed by the holder of parental authority.
* Parents affiliated to a social security scheme
* Parents who to live in cities of Saint-Etienne, Villars, Saint Priest-en-Jarez, Etrat and Saint Jean-Bonnefonds, France

Exclusion Criteria:

* inter-uterine growth restriction
* antenatal neurological pathologies or at birth
* perinatal asphyxial encephalopathy
* antenatal pathologies (e.g. trisomy 21, hydrocephalus...)
* multiple pregnancy

Ages: 1 Day to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants at the birth
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Acoustic structures crying of parameters Principal Component 1 (PC1) and Principal Component 2 (PC2) | up to 3 and half months.
  Comparison of acoustic structures crying of parameters Principal Component 1 (PC1) and Principal Component 2 (PC2) with PRAAT software.

SECONDARY OUTCOMES:
Questionnaire of cry in infant | up to 3 and half months.
  At every cry, parent should answer at the questionnaire of cry in infant: context of the crying (situation), how he interpreted it (pain, hunger, discomfort, etc.), actions he undertook to calm the crying (reassurance, lift, change, breastfeeding), and if those they have been effective in comforting the baby.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MATHEVON, PhD, Study Chair — Université Jean MONNET, Saint-Etienne, France
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No